CLINICAL TRIAL: NCT03587467
Title: Study on Gut Microbiota in Chronic Hepatitis B Virus Infected Patients
Brief Title: Study on Gut Microbiota in Chronic HBV Infected Patients
Acronym: HBV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018001
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Chronic Hepatitis B Infection; Healthy
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- health: 1. Alcohol free history or alcohol consumption <140g per week in male, <70g per week in female
  2. smooth and soft stool like sausage or snake
  3. Voluntary participate in this study
  Interventions: Other: collect fecal specimens
- chronic hepatitis b carrier: 1. Alcohol free history or alcohol consumption <140g per week in male, <70g per week in female
  2. Meet diagnostic criteria of chronic HBV infection in "EASL 2017 Clinical Practice Guidelines on the management"
  Interventions: Other: collect fecal specimens
- chronic hepatitis b: 1. Alcohol free history or alcohol consumption <140g per week in male, <70g per week in female
  2. Meet diagnostic criteria of chronic hepatitis B in "EASL 2017 Clinical Practice Guidelines on the management"
  Interventions: Other: collect fecal specimens
- decompensated cirrhosis: 1. Alcohol free history or alcohol consumption <140g per week in male, <70g per week in female
  2. Meet diagnostic criteria of chronic hepatitis B in "EASL 2017 Clinical Practice Guidelines on the management"
  Interventions: Other: collect fecal specimens

INTERVENTIONS:
Other: collect fecal specimens — collect fresh fecal specimens of participants

SUMMARY:
Hepatitis B Virus(HBV) infection is a common infectious disease affecting up to 2 billion people worldwide. Around 650 thousand people died of liver failure, cirrhosis and primary liver cancer caused by chronic hepatitis B every year. Age is the main factor affecting the chronicity of hepatitis B, while 90% and 25% to 30% of hepatitis b virus(HBV) infection in perinatal and infant period will develop into chronic infection respectively. Whereas the proportion in patients above 5 years old is only 5% to 10%. Intestinal microbiota plays an important role in maintaining nomal physiological function of the intestine and the immune function of the body. It has been found that the disorder of intestinal microbiota is associated with numerous intestinal and parenteral diseases. Recently, the relationship between immune response and intestinal microbiota has been claimed. In a previous study using IMT to treat HBeAg positive chronic hepatits B patients combined with antiviral theraopy, 80% of them has reached HBeAg clearance. Increasing evidence suggests that the gut microbiota has evolved as a new important player in the pathogenesis of hepatitis B virus-induced chronic liver disease. However, the composition and structure alteration of the gut microbiota associated with the stage and progression of HBV infection remains unknown. Hence, we proposed a trial to detected gut microbiota of chronic HBV infected patients high-throughput 16S rRNA gene sequencing to elucidate the microbial influence which contribute to the microbial shift of patient in different stage.

ELIGIBILITY:
Inclusion Criteria:

1. Alcohol free history or alcohol consumption <140g per week in male, <70g per week in female
2. smooth and soft stool like sausage or snake
3. Voluntary participate in this study

Exclusion Criteria:

1. Syptom of digestive system disorder such as hematochezia, constipation, Abdominal distention, abdominal pain, diarrhea and jaundice within 1 month
2. Abormal results of several tests including: fecal routine, fecal occult blood test
3. Be diagnosed as enteritis within 1 month
4. Chronic obstructive pulmonary disease, renal insufficiency and other systemic diseases.
5. Autoimmune disease
6. Chronic fatigue syndrome and neuropsychic disease
7. A history of antibiotics, microecological preparation, gastrointestinal motility medicine, laxative, weight loss drug, Glucose lowering, blood fat regulation, glucocorticoid or immunosuppressor treatment within 1 month
8. History of organic diseases in digestive system such as gastrointestinal polyposis, ulcers, malignancies, etc.
9. History of gastrointestinal surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: chronic hepatitis b virus infected
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota | 1day
  detected gut microbiota of participants through high-throughput 16S rRNA gene sequencing to elucidate the microbial influence which contribute to the microbial shift of patient in different stage.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided